CLINICAL TRIAL: NCT05602506
Title: Safety, Tolerability, and Efficacy of a Dose Reduction Strategy Based on Bictegravir/Emtricitabine/Tenofovir Alafenamide in Virologically Suppressed HIV-infected Adults
Acronym: BETAF-RED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Clinical Professor, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BETAF-RED
Record Dates: First submitted 2022-10-19; First posted 2022-11-02 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- BETAF OD arm (Active Comparator): one tablet taken orally once daily
  Interventions: Drug: Biktarvy 50 mg/200 mg/25 mg film-coated tablets
- BETAF 3W arm (Experimental): one tablet taken orally 3 days per week : Mondays, Wednesdays, and Fridays
  Interventions: Drug: Biktarvy 50 mg/200 mg/25 mg film-coated tablets
- BETAF 2W arm (Experimental): one tablet taken orally 2 days per week : Mondays, and Thursdays
  Interventions: Drug: Biktarvy 50 mg/200 mg/25 mg film-coated tablets
- BETAF 1W arm (Experimental): one tablet taken orally 1 days per week : Mondays
  Interventions: Drug: Biktarvy 50 mg/200 mg/25 mg film-coated tablets

INTERVENTIONS:
Drug: Biktarvy 50 mg/200 mg/25 mg film-coated tablets — The duration of the study treatment will be 48 weeks.

SUMMARY:
This is a phase IV, unicentric, open, pilot, randomized, controlled trial to evaluate Bictegravir/FTC/TAF. The study will be developed at a single clinical care centre:Hospital Clínic de Barcelona, Barcelona, Spain. The aim of this study is to assess the feasibility of dose redutions of Bictegravir/FTC/TAF in virologically suppressed HIV-infected adults on BETAF once daily. The reduction of drug exposure will have a significant positive impact on parameters reflecting potential toxicities associated with bictegravir or tenofovir.

DETAILED DESCRIPTION:
The Primary objectives are:

1. To assess viral efficacy of the reductions of BETAF regimen dose at 12 weeks (on-treatment and intent-to-treat populations).
2. To asess viral efficacy of the reduction of BETAF regimen dose at 48 weeks (on-treatment and intent-to-treat populations).

ELIGIBILITY:
Inclusion Criteria:

* Stable and asymptomatic HIV-infected adults (≥18 years) on BETAF once daily for at least the previous 6 months.
* Plasma HIV-1 RNA less than 50 copies/mL for at least the previous 6 months.
* CD4 cell counts greater than 350 cells/mL at the time of consideration for the study.
* Women of child-bearing potential must have a negative pregnancy test in serum before the inclusion in the study and agree to use highly effective contraceptive methods.
* Patients agreed to participate.

Exclusion Criteria:

* Prior virological failure to any antiretroviral regimen or documented.
* Any diagnosis of psychiatric illness.
* Alcohol abuse or illicit drug consumption (based on their past medical history and specific questions at the time of recruitment).
* Patients co-infected with HIV and active hepatitis B or C virus.
* Any other condition at the doctor's discretion that did not allow ensuring a correct adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Viral efficacy of the reduction of BETAF regimen dose per week at 12 weeks. | at 12 weeks
  standard plasma viral load, lower limit of detection HIV RNA 50 copies/mL
Viral efficacy of the reduction of BETAF regimen dose per week at 48 weeks. | at 48 weeks.
  standard plasma viral load, lower limit of detection HIV RNA 50 copies/mL

SECONDARY OUTCOMES:
Virological efficacy assessed by Standard plasma viral load | at 4, 24, and 36 weeks.
  -Standard plasma viral load, lower limit of detection HIV RNA 50 copies/mL)
Virological efficacy assessed by Blips (VL ≥50 copies/mL followed) | at 0, 4, 12, 24, 36, and 48 weeks
  -Blips (VL ≥50 copies/mL followed)
Virological efficacy assessed by Target not detected with standard plasma viral load (VL ≥ HIV RNA 50 copies/mL) | at 0, 4, 12, 24, 36, and 48 weeks
  -Target not detected with standard plasma viral load (VL ≥ HIV RNA 50 copies/mL)
Virological efficacy assessed by Ultrasensitive plasma viral load (lower limit of detection 5 copies/mL) | at 0, 12, and 48 weeks.
  -Ultrasensitive plasma viral load (lower limit of detection 5 copies/mL)
Virological efficacy assessed by HIV-1 reservoir (total and integrated DNA (copies/106 PBMC)) in CD4 cells | at 0, 12, and 48 weeks.
  - HIV-1 reservoir (total and integrated DNA) in CD4 cells
Virological efficacy assessed by ultra-deep sequencing of plasma and intracellular viral load to detect genotypic resistance | at 0, 4, 12, 24, 36 and 48 weeks
  In case of virological failure, ultra-deep sequencing of plasma and intracellular viral load to detect genotypic resistance
Immunological safety assessed by CD4 and CD8 cells | at 0, 12 and 48 weeks
  -CD4 and CD8 (cells/mL) will be combined to report CD4/CD8 ratio.
Immunological safety 2 assessed by hsCRP, IL-6 and adiponectin levels | at 0, 12 and 48 weeks
  -Inflammation (hsCRP, IL-6, adiponectin) (µg/mL), IL-6 (pg/mL), adiponectin (µg/mL) levels
Immunological safety assessed by sCD14 and CD163 as a Immune activation markers | at 0, 12 and 48 weeks
  - sCD14(ng/l ) and CD163 (ng/l) plasma levels
Subclinical toxicity assessed by BMI index | at 4, 12, 24, 36, and 48
  - Weight and body mass index (BMI)(kg/m2) changes
Body composition assessed by DEXA scan | at 0 and 48 weeks
  -Body composition (g/cm) (fat, fat-free mass, and bone by DEXA)
Impact on sleep quality assessed by Pittsburg Sleep Quality | at 0 and 48 weeks
  - Impact on sleep quality will be evaluated througth Pittsburg Sleep Quality (visual analog score)questionaire at 0 and 48 weeks
Quality of life questionnaire assessed by EuroQol Group EQ-5D™ questionnaire | at 0 and 4,12,24,36, 48 weeks
  - Impact on quality of life will be evaluated througth EuroQol Group EQ-5D™ (Units on a Scale)
Minimum plasma concentration of bictegravir, emtricitabine and tenofovir (Cmim) assessed by Plasma levels of bictegravir, emtricitabine and tenofovir | at 0, 12, and 48 weeks
  - Minimum plasma concentration of bictegravir, emtricitabine and tenofovir (Cmim) (μg/L)
Minimum intracellular concentration of bictegravir, emtricitabine and tenofovir (Cmim) | at 0, 12, and 48 weeks
  Minimum intracellular concentration of bictegravir, emtricitabine and tenofovir (Cmim) (μg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic i Provincial Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No